CLINICAL TRIAL: NCT03290859
Title: Pragmatic Clinical Trial of Race-Specific Response to Propofol Infusion Titrated to Effect for Procedural Sedation During Endoscopy
Brief Title: Race-Specific Propofol Titration to Effect for Procedural Sedation
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201701064 - N; UL1TR001427 (NIH); OCR18882 (Other: University of Florida)
Record Dates: First submitted 2017-09-18; First posted 2017-09-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Unconsciousness; Apnea, Postanesthetic; Sedative Overdose; Hypoxemia
Keywords: Procedural Sedation
MeSH Terms: conditions — Unconsciousness; Butyrylcholinesterase deficiency; Hypoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Compare in buccal samples the frequency of cytochrome allele carrier status in patients exhibiting sensitivity to propofol during the procedural time against published frequency data in Single Nucleotide Polymorphism database (dbSNP) by race.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training intervention: Train anesthesia providers who deliver propofol sedation for GI endoscopy procedures to follow a uniform propofol monotherapy administration guideline to titrate propofol monotherapy infusion to effect according to a standardized protocol.
  Interventions: Procedure: Titrate propofol monotherapy infusion to effect
- Effectiveness of training intervention: Compare the effectiveness of training intervention and standardized titration to effect through aggregate data for metrics of recovery times.

INTERVENTIONS:
Procedure: Titrate propofol monotherapy infusion to effect — Train anesthesia providers in a standardized protocol for titrating propofol infusion to effect.
  Groups: Training intervention

SUMMARY:
Prospectively evaluate newly established guidelines and make clinicians aware of inter-racial difference in propofol sensitivity.

DETAILED DESCRIPTION:
The primary motivation in conducting this study is to conduct the implementation science, i.e., formalize and train, and retrain if needed, anesthesia providers in the standard practice of titrating infusion rate to effect and clinically evaluate the effect of race and ethnicity on propofol monotherapy sedation during GI endoscopy. The ultimate goal is to make it less likely that patients from races known to be sensitive to propofol experience inadvertent overdosing.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing propofol sedation at Gainesville (GNV) and Jacksonville (JAX) GI Endoscopy suites
* Age range 18 - 80 years old
* Patients whose race can be identified from the electronic patient information chart (EPIC)

Exclusion Criteria:

* Patients who identify as multiracial in Epic
* Patients who identify as Other in Epic
* Patients who refuse to indicate their race in Epic
* Patients whose race is listed as unknown in Epic

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing propofol sedation at Gainesville (GNV) and Jacksonville (JAX) GI Endoscopy suites
Sampling Method: Non-Probability Sample
Enrollment: 2780 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-05 (Actual)

PRIMARY OUTCOMES:
Change in the recovery times among races and ethnicities | Change from baseline up to 24 hours
  Monitored using aggregate data for metrics of recovery times

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey White, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No